CLINICAL TRIAL: NCT03353298
Title: A Randomized, Double-blind, Placebo-controlled, 9-month, Parallel Group Study of Allopurinol to Reduce Left Ventricular Mass in Living Kidney Donors (AL-DON)
Brief Title: Lowering Uric Acid in Live Kidney Donors
Acronym: AL-DON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Dag Olav Dahle, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017/397 C; 2017-000666-30 (EudraCT Number)
Record Dates: First submitted 2017-11-10; First posted 2017-11-27 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Renal Transplant Donor of Left Kidney; Renal Transplant Donor of Right Kidney
Keywords: Uric acid; Left ventricular mass; Nephrectomy; Allopurinol; Magnetic resonance imaging
MeSH Terms: interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Allopurinol 300 mg
  Interventions: Drug: Allopurinol 300 mg
- Arm B (Placebo Comparator): Placebo Oral tablets
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Allopurinol 300 mg — Allopurinol oral tablets 300 mg given to participants once daily for 9 months
  Arms: Arm A
Drug: Placebo Oral Tablet — placebo oral tablets given to participants once daily for 9 months
  Arms: Arm B

SUMMARY:
Recently there was described an increase in left ventricular mass after kidney donation. It is uncertain whether this is reversible or not. Allopurinol lowers uric acid in the blood and is normally indicated for gout, but studies have showed that it also can reduce the thickness of the left ventricle of the heart in people with heart- and kidney disease.

The investigators wish to give allopurinol or placebo to kidney donors based on randomization and investigate if this has the same effect on kidney donors. The investigators are assessing this by performing a cardiac MRI at baseline and after 9 months of treatment. In addition the investigators wish to see if allopurinol can have beneficial effects on blood pressure and insulin sensitivity as well.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney donor ≥ 6 months after donor nephrectomy
2. Donor nephrectomy undertaken in Norway
3. Male or female subject ≥ 18 years old
4. eGFR >30 ml/min/1.73 m2
5. Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

1. Adverse reactions to allopurinol or other xanthine oxidase inhibitors
2. Use of uric acid lowering therapy within 3 months
3. History of gout, xanthinuria or other indications for uric acid lowering therapy such as cancer chemotherapy
4. History of renal calculi
5. History of coronary heart disease
6. Heart failure with left ventricular ejection fraction <45%
7. History of significant (i.e. non-physiological) cardiac valvular stenosis or insufficiency
8. History of clinically significant hepatic disease including hepatitis B or C and/or ALAT (SGPT) above the upper reference limit at screening.
9. History of HIV or AIDS
10. Severe systemic infections, current or within the last 6 months
11. History of malignancy other than localized basal cell carcinoma of the skin, treated or untreated, within the past 5 years.
12. Other life-threatening diseases
13. Haemoglobin concentration < 11 g/dL(males), <10 g/dL (females); white blood cell (WBC) count < 3.5 * 10^9/L; platelet count <50 *10^9/L at screening
14. Use of the following medications at or within 14 days before the screening visit: azathioprine, mercaptopurine, vidarabin, chlorpropamide, warfarin, tamoxifen, theophylline, amoxicillin/ampicillin, cyclophosphamide, doksorubicin, bleomycin, prokarbazin, cyclosporine, didanosine.
15. Contraindications to MRI, including: Magnetic intracranial clips. Metal fragments in orbita. Cochlea (ear) implant. Neurostimulator. Pacemaker/ICD or remaining pacemaker electrodes. Harrington rods in thorax. Claustrophobia. Unable to lie supine.
16. Pregnant or nursing (lactating) women
17. Fertile women, unless they are using effective contraception during dosing of study treatment
18. Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass | Nine months
  Measured change in left ventricular mass using Cardiac MRI, comparing from baseline to 9 months of treatment With allopurinol compared to placebo.

SECONDARY OUTCOMES:
Change in blood pressure | Nine months
  Change from baseline to 9 months in the allopurinol group compared to placebo in systolic and diastolic ambulatory blood pressure, systolic and diastolic Office blood pressure.
Estimated insulin sensitivity, metabolic clearance rate of glucose | Nine months
  Change from baseline to 9 months in the allopurinol group compared to placebo in insulin sensitivity using an orgal glucose tolerance test to measure estimated metabolic clearance rate of glucose, insulin sensitivity, firth-phase insulin release and second-phase insulin release.
Number of antihypertensive medications | Nine months
  Change from baseline to 9 months in the allopurinol group compared to placebo in number of antihypertensive medications
Doses of antihypertensive medications | Nine months
  Change from baseline to 9 months in the allopurinol group compared to placebo in doses of antihypertensive medications
Change in urinary albumin excretion | Nine months
  Change from baseline to 9 months in the allopurinol group compared to placebo in urinary albumin excretion by measuring urinary albumin/creatinine ratio.
Change in estimated GFR | Nine months
  Change from baseline to 9 months in the allopurinol group compared to placebo in estimated GFR

CONTACTS AND LOCATIONS:
Overall Officials: Dag Olav Dahle, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moody WE, Ferro CJ, Edwards NC, Chue CD, Lin EL, Taylor RJ, Cockwell P, Steeds RP, Townend JN; CRIB-Donor Study Investigators. Cardiovascular Effects of Unilateral Nephrectomy in Living Kidney Donors. Hypertension. 2016 Feb;67(2):368-77. doi: 10.1161/HYPERTENSIONAHA.115.06608. PMID 26754643
- [Background] Kao MP, Ang DS, Gandy SJ, Nadir MA, Houston JG, Lang CC, Struthers AD. Allopurinol benefits left ventricular mass and endothelial dysfunction in chronic kidney disease. J Am Soc Nephrol. 2011 Jul;22(7):1382-9. doi: 10.1681/ASN.2010111185. Epub 2011 Jun 30. PMID 21719783
- [Background] Altmann U, Boger CA, Farkas S, Mack M, Luchner A, Hamer OW, Zeman F, Debl K, Fellner C, Jungbauer C, Banas B, Buchner S. Effects of Reduced Kidney Function Because of Living Kidney Donation on Left Ventricular Mass. Hypertension. 2017 Feb;69(2):297-303. doi: 10.1161/HYPERTENSIONAHA.116.08175. Epub 2017 Jan 3. PMID 28049698
- [Background] Rekhraj S, Gandy SJ, Szwejkowski BR, Nadir MA, Noman A, Houston JG, Lang CC, George J, Struthers AD. High-dose allopurinol reduces left ventricular mass in patients with ischemic heart disease. J Am Coll Cardiol. 2013 Mar 5;61(9):926-32. doi: 10.1016/j.jacc.2012.09.066. PMID 23449426
- [Background] Szwejkowski BR, Gandy SJ, Rekhraj S, Houston JG, Lang CC, Morris AD, George J, Struthers AD. Allopurinol reduces left ventricular mass in patients with type 2 diabetes and left ventricular hypertrophy. J Am Coll Cardiol. 2013 Dec 17;62(24):2284-93. doi: 10.1016/j.jacc.2013.07.074. Epub 2013 Aug 28. PMID 23994420

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03353298/Prot_SAP_000.pdf